CLINICAL TRIAL: NCT03767439
Title: Trial of Nivolumab With Vismodegib in Patients With Basal Cell Nevus Syndrome (BCNS)
Brief Title: Nivolumab With Vismodegib in Patients With Basal Cell Nevus Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Loss of funding
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Richard D. Carvajal, Assistant Professor of Medicine at the Columbia University Medical, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAS1021
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Basal Cell Nevus Syndrome
Keywords: Nivolumab; Vismodegib; Basal Cell; Basal Cell Nevus Syndrome (BCNS)
MeSH Terms: conditions — Basal Cell Nevus Syndrome | interventions — HhAntag691; Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nivolumab, Vismodegib, Ipilimumab (Experimental): Patients will receive a two week run-in of Vismodegib 150 mg PO daily followed by concurrent Nivolumab 480 mg IV every 4 weeks and Vismodegib 150 mg PO daily.
  In an exploratory fashion, patients will have the option to receive combination Ipilimumab 1 mg/kg IV every 6 weeks and Nivolumab 360 mg IV every 3 weeks at the time of disease progression.
  Interventions: Drug: Vismodegib; Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Vismodegib — 150 mg PO daily
  Other Names: ERIVEDGE
Drug: Nivolumab — 480 mg IV every 4 weeks
  Other Names: OPDIVO
Drug: Ipilimumab — 1 mg/kg IV every 6 weeks
  Other Names: YERVOY

SUMMARY:
This is a single-arm, phase II study to assess the efficacy of combined SMO and PD-1 inhibition with Vismodegib (SMO inhibitor) and Nivolumab (anti-PD-1 antibody) in BCNS patients (target enrollment of 22 patients), with a primary endpoint of 18-month disease control rate. The purpose of this study is to test the hypothesis that Nivolumab and Vismodegib will improve the percentage of BCNS patients who achieve disease control (defined as total tumor burden <50% of baseline) at 18 months from 50% to 80%. Baseline and on-treatment biopsies will be obtained to characterize the immune effects of combined SMO and PD-1 inhibition.

DETAILED DESCRIPTION:
Basal cell carcinoma (BCC) is by far the most common form of human malignancy, affecting more than 3.5 million Americans each year. Aberrant activation of the Hedgehog (Hh) pathway, typically through loss of the receptor Patched (PTCH) or oncogenic activation of Smoothened (SMO), has been identified as the primary driver of BCC growth and development. In particular, up to 1 in 57,000 individuals in the US are affected by a rare, autosomal dominant disorder characterized by mutations in protein patched homolog 1 (PTCH1) known as basal cell nevus syndrome (BCNS). These patients can develop dozens to hundreds of BCCs at any one time (1-5). Surgical removal of the entire tumor burden is not feasible.

Hh-targeted therapies employing inhibitors of SMO (i.e., Vismodegib, Sonidegib) have shown remarkable efficacy in reducing tumor burden in BCC patients. However, the sustained clinical utility of these agents has been hampered by the rapid development of clinical resistance, significant tumor recurrence, and toxicity. Treatment strategies directed at finding additional molecular or immunological targets may enhance the possibility of sustained remission and/or cure of these tumors. Emerging data from our research group and others suggest the therapeutic efficacy of SMO inhibition may be dependent on immunological mechanisms. Hh inhibition appears to increase T cell recruitment and activation as well as upregulate major histocompatibility complex (MHC) class I expression on tumor cells. These data, together with case reports demonstrating the efficacy of cytotoxic T-lymphocyte associated protein 4 (CTLA-4) and programmed death-1 (PD-1) inhibition in Hh inhibitor-naïve and resistant BCCs, support a role for anti-tumor immunity in BCC and underscore the potential enhanced therapeutic efficacy of combined SMO and immunological checkpoint inhibition.

ELIGIBILITY:
Inclusion Criteria:

* 10 or more surgically eligible BCCs (SEBS) within the prior 2 years
* Age > 16 years
* Karnofsky Performance Score (KPS) > 60%, Eastern Cooperative Oncology Group (ECOG) < 2
* Prior SMO inhibitor therapy is permitted, but patients must have developed new and/or progressive lesions on or after therapy
* Adequate organ function
* All clinically significant toxicities from prior systemic therapy must be < Grade 1
* Subjects must agree to undergo four serial tumor biopsies (may be of different tumors) at baseline, after a two week run-in of Vismodegib, between 4-6 weeks of concurrent Nivolumab and Vismodegib, and at the time of disease recurrence or progression.

Exclusion Criteria:

1. Prior therapy with an immunological checkpoint inhibitor
2. Prior SMO inhibitor therapy is permitted, but patients must have developed new and/or progressive lesions on or after therapy
3. Routine use of topical (applied to >5% of skin) or systemic therapies that might interfere with evaluation of the study medication in the prior 4 weeks

   1. Topical corticosteroids
   2. Systemic or topical retinoids e.g., etretinate, isotretinoin, tazarotene, tretinoin, adapalene
   3. Topical alpha-hydroxy acids e.g., glycolic acid, lactic acid
   4. Systemic or topical 5-fluorouracil or imiquimod to skin above the knees
4. Patients who have not recovered from adverse events (> Grade 1) due to prior treatments
5. Treatment with any other investigational agents
6. Recent major surgery within 4 weeks prior to starting study treatment. Minor surgeries such as placement of vascular access are not exclusionary.
7. Known history of hypersensitivity to any of the ingredients in the study medication formulations
8. Requirement for immunosuppressive corticosteroids at doses exceeding 10 mg prednisone daily or equivalent prior to first dose of Nivolumab
9. Ongoing or recent (within 5 years) evidence of significant autoimmune disease at baseline or associated with prior therapy requiring treatment with systemic immunosuppressive treatments with the exception of:

   1. Viligo
   2. Childhood asthma that has resolved
   3. Residual endocrinopathies requiring replacement therapy
   4. Psoriasis that does not require systemic treatment
10. History of solid organ transplant
11. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
12. Uncontrolled hypocalcemia, hypomagnesemia, or hypokalemia
13. HIV positive patients on combination antiretroviral therapy
14. Refractory nausea and vomiting, active gastrointestinal disease e.g. inflammatory bowel disease, or significant bowel resection that would preclude adequate absorption
15. Have evidence of any other significant skin condition, clinical disorder, physical examination finding, or laboratory finding that, as judged by the investigator, makes it undesirable for the patient to participate in the study
16. Active treatment for a second malignancy
17. Pregnant women are excluded from this study because nivolumab, ipilimumab and vismodegib may be teratogenic or have abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with nivolumab, ipilimumab or vismodegib, breastfeeding should be discontinued if the mother is receiving study treatment.
18. Male patients unwilling or unable to comply with pregnancy prevention measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Disease control rate | 18 months
  Defined as the percentage of patients achieving a total tumor burden <50% of baseline tumor burden

SECONDARY OUTCOMES:
Total Number of Adverse Reactions | 18 months
  Testing safety and toxicity assessed using CTCAE v5.0 criteria
Disease Control Rate (DCR) | 18 months
  DCR is defined as the percentage of subjects who have achieved complete response (CR), partial response (PR), or stable disease (SD) based on assessments per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Duration of Response (DOR) | 18 months
  For subjects who demonstrate CR or PR, based on assessments per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Carvajal, MD., Principal Investigator — Columbia University